CLINICAL TRIAL: NCT06598020
Title: Evaluating the Impact of an Integrative Oncology Training Program for Physicians, Nurses, and Medical Educators on Knowledge, Attitudes, and Implementation of Learned Clinical Skills
Brief Title: Evaluating the Impact of an Integrative Oncology Training Program for Healthcare Providers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Collaborators: Advot Fund of Reality Group (Unknown); Israel Cancer Association (Other)
Responsible Party: Principal Investigator, Eran Ben-Arye, Director, Integrative Oncology Program, Lin Medical Center, Technion, Israel Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TEC-050623
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Integrative Oncology; Medical Education; Palliative Care
Keywords: Medical education; Integrative oncology; Oncology; Supportive care
MeSH Terms: conditions — Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced competency curriculum-based training (Experimental): Trainees allocated to this arm undergo practical training, based on the five-item competency curriculum adapted from the list of knowledge, skills, and ability-related competencies recommended by the Society for Integrative Oncology.
  Interventions: Behavioral: Supportive Care
- Standard training arm (Experimental): Trainees in this arm will observe from the side practitioner-patient interaction in integrative oncology setting of care
  Interventions: Behavioral: Supportive Care

INTERVENTIONS:
Behavioral: Supportive Care — Competency-based training purposed to alleviate anxiety relief using a mind-body modality and improve pain with touch modalities (e.g., acupressure)

SUMMARY:
The goal of this study is to learn about the short- and long-term effects of two medical education approaches to teaching integrative oncology (IO) in a multi-disciplinary group of healthcare providers attending a national IO training. The main question it aims to answer is: Does active medical education approach focusing on IO-related skills is associated with better training outcomes compared to clerkship-based observation of IO clinics? Participants (trainees) will answer online survey questions about their knowledge, attitudes, and clinical proficiencies along the training process.

DETAILED DESCRIPTION:
The study is conducted within a multi-centered, prospective, controlled and randomized format, using a mixed quantitative and qualitative methodology. Participants eligible for study inclusion are healthcare providers (HCPs, nurses, physicians, para-medical, or complementary medicine practitioners), age ≥ 18 years enrolling in a structured IO training program. Trainees are randomly allocated to either the Enhanced IO Training arm (Group A) or Standard IO Training arm of the study (Group B). Participants in both study arms undergo 110-hour online section of the IO training course, followed by 170-hour practical training.

Those in the Enhanced IO Training arm undergo practical training, based on the five-item competency curriculum adapted from the list of knowledge, skills, and ability-related competencies recommended by the Society for Integrative Oncology. The five-item competency-based curriculum include the following two clinical implementation competencies:

* Anxiety relief using a mind-body modality (e.g., breathing, relaxation, guided imagery)
* Improving pain with touch modalities (e.g., acupressure, acupuncture, reflexology), including use of acupressure points with established effectiveness in the reduction of cancer pain Participants in the Standard IO training group (Group B) will observe from the side during the IO practitioner-patient interaction.

The practical section of the training program will include two mentoring days, the first scheduled at the beginning of the 110-hour theory-based IO training, the second at the conclusion of this training. Participants in both study groups will be exposed during the two mentoring days to between 3-5 clinical IO therapeutic interactions with patients admitted to the oncology center.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare providers (nurses, physicians, para-medical, or complementary medicine practitioners) who have applied to and been accepted for the integrative oncology training program

Exclusion Criteria:

* Healthcare providers who were not received a letter of support from the medical administrator stating commitment to allocate at least 5 hours weekly post-training to enable the trainee practicing integrative oncology care in the medical center.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Integrative oncology competency assessment | At each of the two assessment points, competencies will be assessed at the beginning of the training and 6 hours later.
  Integrative oncology clinical competencies will be assessed while scoring five-item competency list provided (knowledge, skill, ability, and two clinical implementation-related competencies), using a visual analogue scale ranging between 1 (very low) and 5 (very high). Competencies will be assessed at two assessment points: 1. At the beginning of the training; 2. Following 9 months, following conclusion of the training.

SECONDARY OUTCOMES:
Qualitative assessment of trainees narratives | 18 months
  Qualitative assessment of trainees' narrative reflections will include open questions on their perspectives regarding any changes they experienced in their knowledge, skills, and ability-related competencies regarding integrative oncology. Qualitative analysis of the trainees' narratives will be conducted using ATLAS.ti software for systematic coding.

CONTACTS AND LOCATIONS:
Overall Officials: Eran Ben-Arye, MD, Principal Investigator — Carmel Medical Center
Locations (1):
- Lin Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Undecided at this point

REFERENCES:
- [Background] Witt CM, Balneaves LG, Carlson LE, Cohen M, Deng G, Fouladbakhsh JM, Kinney AY, Mehta A, Mailman J, Pole L, Rogge AA, O'Toole C, Zick SM, Helmer SM. Education Competencies for Integrative Oncology-Results of a Systematic Review and an International and Interprofessional Consensus Procedure. J Cancer Educ. 2022 Jun;37(3):499-507. doi: 10.1007/s13187-020-01829-8. PMID 32783117